CLINICAL TRIAL: NCT01340456
Title: Induction of Drug Metabolism by Rifampicin to Compare the Endogenous Biomarker 4beta-OHcholesterol With the Probe Drug Midazolam as Quantitative Markers for Cytochrome P450 3A4 Induction
Brief Title: Cholesterol Metabolites as Markers for CYP3A Induction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Tobias Bäckström, Department of Clinical Pharmacology, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1001-01
Record Dates: First submitted 2011-04-15; First posted 2011-04-22 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-05

CONDITIONS: CYP3A4 Induction
Keywords: 4beta-OHcholesterol; Midazolam; CYP3A4; Enzyme induction; Drug metabolism
MeSH Terms: interventions — Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rifampicin 10 mg QD (Experimental)
  Interventions: Drug: Rifampicin treatment
- Rifampicin 20 mg QD (Experimental)
  Interventions: Drug: Rifampicin treatment
- Rifampicin 100 mg QD (Experimental)
  Interventions: Drug: Rifampicin treatment

INTERVENTIONS:
Drug: Rifampicin treatment — induction of CYP3A4 with one of three rifampicin doses (10, 20, 100 mg QD)
  Other Names: Rifadin

SUMMARY:
The objectives of this study are:

* To investigate if the endogenous cholesterol metabolite, 4beta-OHcholesterol could be used as a marker for induction of cytochrome P450 (CYP) 3A4.
* To compare 4beta-OHcholesterol with midazolam as a marker for induction of CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

1. Females and males.
2. Age of 18 and above.
3. Caucasians.
4. Healthy as assessed by medical history and examination by principal investigator or delegated personnel.
5. Accept to refrain from herbal drugs, natural preparations, and grapefruit juice 48 hours before and during the study period.
6. Accept to completely refrain from alcohol during day -1 to 1 and R14-R16. During the rest of the study moderate alcohol use is permitted (equal to 1 glass of wine or 1 beer per day).
7. Women of childbearing age should accept using a reliable barrier contraceptive method throughout the study.
8. Women of childbearing age should have a negative pregnancy test at the screening visit.
9. Capable of following given instructions.
10. Has given written informed consent after receiving both oral and written study information.

Exclusion Criteria:

1. Predisposal to allergic drug reactions.
2. Anamnestic and/or visual signs of infection.
3. Women are not allowed to use oral hormone-based contraceptives 2 weeks before start of study and during the study.
4. Participation in another study within one month before entering the present study.
5. Intake of any other drug that can influence the enzyme activity of CYP3A4.
6. Pregnancy.
7. Breast-feeding.
8. A history of liver disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Change in 4beta-OHcholesterol | Directly before treatment with rifampicin and 14 days after the end of treatment with rifampicin
  The primary objective of the study is to investigate whether the endogenous cholesterol metabolite 4β-hydroxycholesterol could be used as a marker for induction of CYP3A4. For this purpose the induction of 4β-hydroxycholesterol formation will be compared to the induction of quinine and midazolam metabolism.

SECONDARY OUTCOMES:
Ratio between midazolam AUC induced and midazolam AUC uninduced | Before treatment with rifampicin and after 14 days of treatment with rifampicin
  Secondary aim of the study is to compare 4β-hydroxycholesterol as a biomarker for CYP3A4 compared to 6β-hydroxycortisol/cortisol ratio, which sometimes is used as a marker for CYP3A4 induction.
  Another secondary aim is to relate our estimations of CYP3A4-expression to measured levels of 25-OH-vitamin D.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Bäckström, MD PhD, Principal Investigator — Department of Clinical Pharmacology, Karolinska University Hospital
Locations (1):
- Clinical Pharmacology Trial Unit (CPTU), Karolinska University Hospital, Stockholm, Sweden